CLINICAL TRIAL: NCT06338969
Title: The Impact of Different Carbohydrate Restriction After a Gastric Bypass on the Manifestation of Starvation Ketosis and Ketoacidosis in Patients With Nonalcoholic Steatohepatitis
Brief Title: The Impact of Different Carbohydrate Restriction After a Gastric Bypass on the Ketosis and Ketoacidosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Society of Bariatric and Metabolic Surgeons of Kazakhstan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PostBariKetosis
Record Dates: First submitted 2024-03-24; First posted 2024-04-01 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Obesity, Morbid; NASH; Ketosis; Keto Acidosis; Carbohydrate Metabolism Disorder
Keywords: Carbohydrate restriction; Ketosis after bariatric surgery
MeSH Terms: conditions — Obesity, Morbid; Ketosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Carbohydrate Restriction after a Gastric Bypass: 51-75% deficit in carbohydrates (Experimental): In the postoperative period, the amount of carbohydrate intake was reduced by counting carbohydrates in a glucose solution in the first three days after surgery and counting carbohydrates in food. Created a carbohydrate deficit of 51-75%.
  Interventions: Other: Carbohydrate Restriction after a Gastric Bypass
- Carbohydrate Restriction after a Gastric Bypass: 26-50% deficit in carbohydrates (Active Comparator): In the postoperative period, the amount of carbohydrate intake was reduced by counting carbohydrates in a glucose solution in the first three days after surgery and counting carbohydrates in food. Created a carbohydrate deficit: 26-50% deficit in carbohydrates.
  Interventions: Other: Carbohydrate Restriction after a Gastric Bypass
- Carbohydrate Restriction after a Gastric Bypass:1-25% deficit in carbohydrates (Active Comparator): In the postoperative period, the amount of carbohydrate intake was reduced by counting carbohydrates in a glucose solution in the first three days after surgery and counting carbohydrates in food. Created a carbohydrate deficit:1-25% deficit in carbohydrates.
  Interventions: Other: Carbohydrate Restriction after a Gastric Bypass

INTERVENTIONS:
Other: Carbohydrate Restriction after a Gastric Bypass — All patients will undergo laparoscopic one anastomotic gastric bypass. In the postoperative period, all patients will receive normal daily amounts of protein and fat. Depending on the amount of carbohydrates that will be received after surgery, patients will randomly (no mask) be divided into three groups:
  The first group: 51-75% deficit in carbohydrates Second group: 26-50% deficit in carbohydrates The third group: has a 1-25% deficit in carbohydrates.
  Other Names: laparoscopic one anastomotic gastric bypass

SUMMARY:
Background:

Ketosis after bariatric surgery is a metabolic process that occurs when the body breaks down fat for energy because of not getting enough carbohydrates.

Insufficient production of ketone bodies reduces the rate of weight loss, and excessive amounts of ketones can lead to ketoacidosis or liver failure in patients with nonalcoholic steatohepatitis (NASH).

The investigators hypothesize that weight loss is directly related to calorie intake, and a significant reduction in carbohydrate content leads to increased ketosis and the risk of ketoacidosis.

Objectives:

The study aimed to compare the incidence of ketoacidosis and liver failure in patients with NASH with different intakes of carbohydrates in the early postoperative period after gastric bypass. In addition, the investigators want to find out how carbohydrate restriction will affect weight loss for up to 1 year.

DETAILED DESCRIPTION:
Methods:

This study is a three-arm randomized controlled trial. All patients will undergo laparoscopic one anastomotic gastric bypass. In the postoperative period, all patients will receive normal daily amounts of protein and fat. Depending on the amount of carbohydrates that will be received after surgery, patients will randomly (no mask) be divided into three groups:

The first group: 51-75% deficit in carbohydrates Second group: 26-50% deficit in carbohydrates The third group: has a 1-25% deficit in carbohydrates.

Primary outcome measurement Compare the incidence of ketoacidosis and liver failure in three groups of patients with NASH with different intakes of carbohydrates in the early postoperative period after gastric bypass.

Secondary outcome measurements Change in body mass index (Δ BMI). Effect weight loss for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* obesity patients BMI 30-50 kg/m2.
* patients with nonalcoholic steatohepatitis (NASH).

Exclusion Criteria:

* patients with active physical sports
* diabetes
* cirrhosis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Cases of ketosis and incidence of ketoacidosis | The time frame is baseline, first 7 days, 1, 3, 6,12 months after surgery.
  Compare the incidence of ketoacidosis and liver failure in three groups of patients with NASH with different intakes of carbohydrates in the early postoperative period after gastric bypass
Cases of liver failure | The time frame is baseline, first 7 days, 1, 3, 6,12 months after surgery.
  Compare the incidence of liver failure in three groups of patients with NASH with different intakes of carbohydrates in the early postoperative period after gastric bypass

SECONDARY OUTCOMES:
Change in body mass index (Δ BMI) | The time frame is baseline,1, 3, 6,12 months after surgery.
  This measurement assesses the change in BMI after the intervention. Weight (kg) and height (cm) will be combined in the BMI (kg/m2).

CONTACTS AND LOCATIONS:
Overall Officials: Oral Ospanov, PhD, Principal Investigator — The Society of Bariatric and Metabolic Surgeons of Kazakhstan
Locations (1):
- Oral Ospanov, Astana, Aqmola, Kazakhstan

IPD SHARING:
Plan to Share IPD: No